CLINICAL TRIAL: NCT00760292
Title: Genetic Variants and Phenotypic Characteristics of Patients With T2DM
Acronym: GenVarT2DM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Danish PhD schools of Molecular Metabolism and Endocrinology (Other); University of Southern Denmark (Other)
Other Study IDs: 034
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Genetic Variants; SNP; DNA microarray
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Type 2 Diabetic Patients
- 2: Non-diabetic individuals

SUMMARY:
Background: Genetic risk-markers associated with T2DM are thoroughly studied. So far, only a few genetic variants, also termed single nucleotide polymorphisms (SNP's), have been replicated in several studies and each of them gives only limited explanation for the growing incidence of T2DM. The hypothesis of the present study is that determination of combinations of genetic variants by SNP-chip technology may improve the prediction of T2DM, complications and efficacy of treatment compared to the methods previously used including genome wide association (GWA) studies. The SNP-chip/ DNA microarray makes it possible to study several SNP's association with T2DM, one by one but also in combination.

Aims: To study whether specific genetic variants, and combinations of these, 1) are present with higher prevalence in patients with T2DM than in the normal population, 2) are associated with specific diabetes-related complications and 3) the effect of the anti-diabetic treatment.

Methods: During the next three years 1000 patients with T2DM and 1000 healthy, non-diabetic persons will be included in the study, and examined by blood samples, a questionnaire and clinical evaluation, all in one visit. Initially, we will perform DNA analyses on blood samples from 372 patients included in another clinical study from our department. Description of genetics will be done by a DNA-chip with approximately 70 SNP's, which have previously been reported to be associated with T2DM.

Results and conclusions: It is expected that the result of this project can help us predicting T2DM, diabetes-related complications and individualizing treatment to the individual patient with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* > 18 years and

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Diabetic Patients from Dept. of Endocrinology, Odense University Hospital
  2. Non-diabetic volunteers found from advertising at Odense University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Endocrinology, Odense University Hospital, Odense, Funen, Denmark